CLINICAL TRIAL: NCT02751775
Title: Physical Activity and Screen-Time Regulations in Childcare Centers: Influence on Young Children's Health Behaviors (Pause & Play) - Aim 3
Brief Title: Physical Activity and Screen-Time Regulations in Childcare Centers - Aim 3
Acronym: Pause and Play
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Amanda Staiano, PBRC Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2015-045; U54MD008602-P02UAB (Other Grant/Funding Number: UAB); U54MD008602 (NIH)
Record Dates: First submitted 2016-04-19; First posted 2016-04-26 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Childhood Obesity
Keywords: Childcare center regulations; Physical Activity; Sedentary Behavior; Screen-Time Behavior; Focus groups
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective is to establish community priorities for strategies to improve young children's health behaviors based on focus groups of stakeholders in the greater Baton Rouge area.

DETAILED DESCRIPTION:
Pause and Play (Aim 3) objective will be achieved through a series of taskforce and focus group meetings administered by the Mayor's Healthy City Initiative (MHCI). Meetings will include monthly meetings of the MHCI advisory boards composed of community stakeholders and focus groups of childcare center directors and parents. Stakeholders will create dissemination and implementation plans to leverage the findings of the project. We plan to conduct 2-3 focus groups of 8-10 parents and childcare directors, for a total of 16-30 participants. Participation in the focus group part of the study will last approximately 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Either a director of a licensed childcare center in East Baton Rouge Parish OR a legal guardian and/or primary caretaker of a child aged 3 to 5 years who is enrolled in a licensed childcare center
* Able to understand and speak English
* Willing to be audio-taped during the focus group (for transcription purposes)

Exclusion Criteria:

* Being affiliated with 1 of the 10 childcare centers being assessed for Pause and Play Aims 1 or 2, either as a director/teacher or as a parent of a student
* Cognitive impairments that interfere with participation in a group discussion

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population will include parents and childcare directors.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Qualitative Concepts, Themes and Quotes of focus group participants | 6 months
  Generation of key words, phrases, and quotes coded as variable themes agreed upon by at least one other participant in the group and repeated independently in other focus groups. Transcripts will be imported into NVivo software (Version 10, QSR, Victoria, Austrailia) to allow for thematic evaluation. The evaluation process will include the following: 1) generation of key words, phrases, and quotes coded as variable themes agreed upon by at least one other participant in the group and repeated independently in another focus group; 2) grouping of variables based on unifying concepts and themes; and 3) review of the variable groupings to ensure consistency and relevance of proposed unifying concepts.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Staiano, PhD, Principal Investigator — PBRC Assistant Professor
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Joseph ED, Kracht CL, St Romain J, Allen AT, Barbaree C, Martin CK, Staiano AE. Young Children's Screen Time and Physical Activity: Perspectives of Parents and Early Care and Education Center Providers. Glob Pediatr Health. 2019 Jul 24;6:2333794X19865856. doi: 10.1177/2333794X19865856. eCollection 2019. PMID 31384633
- [Result] Staiano AE, Allen AT, Fowler W, Gustat J, Kepper MM, Lewis L, Martin CK, Romain JS, Webster EK. State Licensing Regulations on Screen Time in Childcare Centers: An Impetus for Participatory Action Research. Prog Community Health Partnersh. 2018;12(1S):101-109. doi: 10.1353/cpr.2018.0025. PMID 29755053
- [Result] Kracht CL, Webster EK, Staiano AE. A natural experiment of state-level physical activity and screen-time policy changes early childhood education (ECE) centers and child physical activity. BMC Public Health. 2020 Mar 24;20(1):387. doi: 10.1186/s12889-020-08533-8. PMID 32209069
- [Result] Webster EK, Martin CK, Staiano AE. Fundamental motor skills, screen-time, and physical activity in preschoolers. J Sport Health Sci. 2019 Mar;8(2):114-121. doi: 10.1016/j.jshs.2018.11.006. Epub 2018 Nov 24. PMID 30997257
- [Result] Staiano AE, Webster EK, Allen AT, Jarrell AR, Martin CK. Screen-Time Policies and Practices in Early Care and Education Centers in Relationship to Child Physical Activity. Child Obes. 2018 Aug/Sep;14(6):341-348. doi: 10.1089/chi.2018.0078. PMID 30199286
- [Result] Martins, C., Webster, E. K., Bandeira, P. F. R., & Staiano, A. E. (2022). Identifying Fundamental Motor Skills Building Blocks in Preschool Children From Brazil and the United States: A Network Analysis. Journal of Motor Learning and Development, 10(1), 96-115. Retrieved Mar 27, 2024, from https://doi.org/10.1123/jmld.2021-0022
- [Result] Kracht CL, Webster EK, Staiano AE. Relationship between the 24-Hour Movement Guidelines and fundamental motor skills in preschoolers. J Sci Med Sport. 2020 Dec;23(12):1185-1190. doi: 10.1016/j.jsams.2020.06.021. Epub 2020 Jul 5. PMID 32653249
- [Result] Kracht CL, Webster EK, Staiano AE. Sociodemographic Differences in Young Children Meeting 24-Hour Movement Guidelines. J Phys Act Health. 2019 Oct 1;16(10):908-915. doi: 10.1123/jpah.2019-0018. Epub 2019 Sep 6. PMID 31491748

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT02751775/Prot_SAP_000.pdf